CLINICAL TRIAL: NCT00005578
Title: Advanced Stage Hodgkins Disease - A Pediatric Oncology Group Phase III Study
Brief Title: Combination Chemotherapy With or Without Dexrazoxane in Treating Children With Hodgkin's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 9425; COG-9425 (Other: Children's Oncology Group); CDR0000065359 (Other: Clinical Trials.gov); P9425 (Other: Pediatric Oncology Group)
Record Dates: First submitted 2000-05-02; First posted 2004-05-26 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Cardiac Toxicity; Lymphoma
Keywords: stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; cardiac toxicity
MeSH Terms: conditions — Cardiotoxicity; Lymphoma | interventions — Bleomycin; Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; Dexrazoxane; Razoxane; Doxorubicin; Etoposide; Prednisone; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Patients are randomized to one of two treatment arms. All patients receive 3 courses of chemotherapy consisting of doxorubicin hydrochloride and etoposide on days 0 and 1, bleomycin sulfate and vincristine sulfate on days 0 and 7, cyclophosphamide on day 0, and prednisone on days 0-6. Filgrastim (G-CSF) is administered on days 5-6 and 8-19. Each course is 21 days in length. Patients assigned to arm I receive only these drugs.
  Interventions: Biological: bleomycin sulfate; Biological: filgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy
- Arm 2 (Experimental): Patients are randomized to one of two treatment arms. All patients receive 3 courses of chemotherapy consisting of doxorubicin hydrochloride and etoposide on days 0 and 1, bleomycin sulfate and vincristine sulfate on days 0 and 7, cyclophosphamide on day 0, and prednisone on days 0-6. Filgrastim (G-CSF) is administered on days 5-6 and 8-19. Each course is 21 days in length. Dexrazoxane hydrochloride on days 0, 1, and 7
  Interventions: Biological: bleomycin sulfate; Biological: filgrastim; Drug: cyclophosphamide; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Biological: bleomycin sulfate
  Other Names: Blenoxane; NSC #125066
Biological: filgrastim
  Other Names: GRANULOCYTE-COLONY STIMULATING FACTOR; r-metHuG-CSF; G-CSF; Neupogen; NSC #614629
Drug: cyclophosphamide
  Other Names: CTX; Cytoxan; NSC #26271
Drug: dexrazoxane hydrochloride
  Other Names: DZR; ADR-529; ZINECARD; ICRF-187; NSC #169780
  Arms: Arm 2
Drug: doxorubicin hydrochloride
  Other Names: Adriamycin; NSC #123127
Drug: etoposide
  Other Names: VP-16; VePesid; NSC #141540
Drug: prednisone
  Other Names: Deltasone; Meticorten; Liquid Pred; NSC #10023
Drug: vincristine sulfate
  Other Names: VCR; Oncovin; NSC #67574
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs, such as dexrazoxane, may protect normal cells from the side effects of chemotherapy.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without dexrazoxane in treating children who have Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of doxorubicin, bleomycin, vincristine, etoposide, prednisone and cyclophosphamide (DBVE-PC) with filgrastim (G-CSF) followed by consolidative radiotherapy in children with advanced stage Hodgkin's disease. II. Tailor therapy based on rapidity of response in order to minimize cumulative drug dosages. III. Compare the efficacy of dexrazoxane in reducing pulmonary and cardiac toxicity of DBVE-based therapy without compromising response.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms. All patients receive 3 courses of chemotherapy consisting of doxorubicin and etoposide on days 0 and 1, bleomycin and vincristine on days 0 and 7, cyclophosphamide on day 0, and prednisone on days 0-6. Filgrastim (G-CSF) is administered on days 5-6 and 8-19. Each course is 21 days in length. Patients assigned to arm I receive only these drugs. Patients assigned to arm II receive dexrazoxane on days 0, 1, and 7 in addition to therapy as in arm I. Patients who exhibit a complete remission (CR) or provisional CR then receive radiotherapy to the regional field 5 days a week for 2.8 weeks. If the disease is not responsive, 2 more courses of chemotherapy are given. Patients whose disease remains nonresponsive or progresses go off the study. Radiotherapy may follow for others. Patients are followed every 3 months for the first year, every 4 months for the second year, every 6 months for the third year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 277 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven Hodgkin's disease of the following stages: Stages IIB, IIIB or IV

PATIENT CHARACTERISTICS: Age: 21 or under Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 2 times upper normal limit Renal: Not specified Other: Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: No prior chemotherapy Endocrine therapy: Less than one week of steroids for management of airway complications Radiotherapy: No prior radiotherapy except emergency radiation to the mediastinum Surgery: Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 219 (Actual)
Dates: Start 1997-03; Primary Completion 2004-10 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Diffusing capacity of the lungs for carbon monoxide (DLCO) | One year post therapy
  The Wilcoxon test will be used to evaluate whether DLCO values differ between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Schwartz, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (63):
- United States (57):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - CCOP - Florida Pediatric, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Memorial Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - MBCCOP - South Texas Pediatric, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - McMaster Division, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
- Swiss Pediatric Oncology Group Bern, Bern, Switzerland

REFERENCES:
- [Background] Tebbi CK, London WB, Friedman D, Villaluna D, De Alarcon PA, Constine LS, Mendenhall NP, Sposto R, Chauvenet A, Schwartz CL. Dexrazoxane-associated risk for acute myeloid leukemia/myelodysplastic syndrome and other secondary malignancies in pediatric Hodgkin's disease. J Clin Oncol. 2007 Feb 10;25(5):493-500. doi: 10.1200/JCO.2005.02.3879. PMID 17290056
- [Background] Schwartz CL, Tebbi CK, Constine LS: Response based therapy for pediatric Hodgkin's disease (HD): Pediatric Oncology Group (POG) protocols 9425/9426. [Abstract] Med Pediatr Oncol 37 (3): A-P219, 263, 2001.
- [Result] Voss SD, Chen L, Constine LS, Chauvenet A, Fitzgerald TJ, Kaste SC, Slovis T, Schwartz CL. Surveillance computed tomography imaging and detection of relapse in intermediate- and advanced-stage pediatric Hodgkin's lymphoma: a report from the Children's Oncology Group. J Clin Oncol. 2012 Jul 20;30(21):2635-40. doi: 10.1200/JCO.2011.40.7841. Epub 2012 Jun 11. PMID 22689804
- [Result] Schwartz CL, Constine LS, Villaluna D, London WB, Hutchison RE, Sposto R, Lipshultz SE, Turner CS, deAlarcon PA, Chauvenet A. A risk-adapted, response-based approach using ABVE-PC for children and adolescents with intermediate- and high-risk Hodgkin lymphoma: the results of P9425. Blood. 2009 Sep 3;114(10):2051-9. doi: 10.1182/blood-2008-10-184143. Epub 2009 Jul 7. PMID 19584400
- [Result] Constine LS, Marcus R, Chauvenet A, et al.: Patterns of failure after response-based, dose-dense therapy for intermediate/high risk pediatric Hodgkin's disease (POG 9425). [Abstract] Int J Radiat Oncol Biol Phys 63 (Suppl 1): A-37, S21, 2005.
- [Result] Schwartz CL, Constine LS, London W, et al.: POG 9425: response-based, intensively timed therapy for intermediate/high stage (IS/HS) pediatric Hodgkin's disease. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1555, 2002.